CLINICAL TRIAL: NCT01020552
Title: ESD: Integrated Services for Women Seeking Postabortion Care in Kenya
Brief Title: Integrating Family Planning Into Postabortion Care
Status: Completed | Type: Observational
Sponsor: FHI 360 (Other)
Collaborators: Pathfinder International (Industry)
Responsible Party: Cate Lane Senior Youth Health Advisor, Pathfinder International
Other Study IDs: 10035
Record Dates: First submitted 2009-11-18; First posted 2009-11-25 (Estimated); Last update posted 2010-04-29 (Estimated); Status verified 2010-04

CONDITIONS: Postabortion Care
Keywords: APHIA II; AIDS, Population, and Health Integrated Assistance project; DCF; data collection forms; FDA; Federal Drug Administration; FP; family planning; IRB; Institutional Review Board; PAC; postabortion care; To document the ESD PAC svc pkg including the provision of services, client satisfaction with those services and provider attitudes towards PAC services; To examine any differences in implementation of the ESD PAC services package for youth and adult clients; To assess the usefulness of five Youth-Friendly PAC Job Aids developed by ESD
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Provision of PAC job aids and provider training on the use of the job aids — Facility-level intervention applied to all study facilities

SUMMARY:
A descriptive post-intervention study designed to provide data to decision-makers at the Kenyan Ministry of Health, the Extending Service Delivery Project (ESD), and Pathfinder International about whether and how to scale-up the ESD Project's postabortion care (PAC) services package. Approximately three months of data will be collected following the introduction of postabortion care job aids in eight public sector health facilities in Central Province and Nairobi, Kenya. Postabortion clients and providers will be interviewed; facilities providing PAC services will be inventoried using facility checklists.

DETAILED DESCRIPTION:
A descriptive post-intervention study designed to provide data to decision-makers at the Kenyan Ministry of Health, the Extending Service Delivery Project (ESD), and Pathfinder International about whether and how to scale-up the ESD Project's postabortion care (PAC) services package. Approximately three months of data will be collected following the introduction of postabortion care job aids in eight public sector health facilities in Central Province and Nairobi, Kenya. Postabortion clients and providers will be interviewed; facilities providing PAC services will be inventoried using facility checklists.

ELIGIBILITY:
Inclusion Criteria:

* For Facilities: APHIA II facilities supported by the ESD project in Central Province and Nairobi, Kenya where: (1) PAC services are provided, (2) at least one provider has received PAC and Youth-friendly PAC training, (3) Community mobilization has been initiated, (4) PAC equipment and supplies have been procured, (5) PAC job aids have been distributed.
* For Clients: Women aged 15 years or older who have received PAC services at a study facility and who have a telephone on which they can be contacted
* For Providers: Any person who offers PAC services at a study facility

Min Age: 15 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: non healthy participants
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2009-09; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Knowledge, attitudes, and practice regarding PAC job aids (clients and providers) | Anticipated end of data collection 12/31/09

SECONDARY OUTCOMES:
Client-report of provider counseling, by client age | Anticipated end of analysis/report writing 4/28/10

CONTACTS AND LOCATIONS:
Overall Officials: Emily Evens, MPH, Principal Investigator — FHI 360; Rose Otieno-Masaba, MD, Principal Investigator — Family Health International - Nairobi
Locations (8):
- Kenya (8):
  - Gatundu District Hospital, Gatundu, Central
  - Karatina District Hospital, Karatina, Central
  - Kerugoya District Hospital, Kerugoya, Central
  - Muranga District Hospital, Muranga, Central
  - Thika District Hospital, Thika, Central
  - Tigoni District Hospital, Tigoni, Central
  - Muthethania Maternity, Nairobi, Nairobi-West
  - Mbagathi District Hospital, Nairobi, West